CLINICAL TRIAL: NCT01757184
Title: A Multicenter, Randomized, Placebo-controlled Study of SBC-102 in Patients With Lysosomal Acid Lipase Deficiency
Brief Title: Acid Lipase Replacement Investigating Safety and Efficacy (ARISE) in Participants With Lysosomal Acid Lipase Deficiency
Acronym: ARISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAL-CL02
Record Dates: First submitted 2012-12-17; First posted 2012-12-28 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Lysosomal Acid Lipase Deficiency
Keywords: Enzyme replacement therapy (ERT); Lysosomal storage disease; Late-onset lysosomal acid lipase deficiency (LAL-D); Acid cholesteryl ester hydrolase deficiency, type 2; Acid lipase disease; Cholesterol ester hydrolase deficiency; LAL-D; LIPA deficiency; Wolman disease; Cholesterol ester storage disease (CESD)
MeSH Terms: conditions — Wolman Disease; Lysosomal Storage Diseases; Cholesterol Ester Storage Disease | interventions — Sebelipase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Double-blind Sebelipase Alfa (Experimental): Double-blind Period: IV infusions of sebelipase alfa at a dose of 1 mg/kg administered qow for 20 weeks.
  Interventions: Drug: Sebelipase Alfa
- Double-blind Placebo (Placebo Comparator): Double-blind Period: IV infusions of matched placebo administered qow for 20 weeks.
  Interventions: Drug: Placebo
- Open-label Sebelipase Alfa/Sebelipase Alfa (Experimental): Participants who were randomized to receive sebelipase alfa during the Double-blind Period and received sebelipase alfa in the Open-label Period. All participants received sebelipase alfa at a dose of 1 mg/kg qow, irrespective of treatment received in the Double-blind Period. Dose modifications were permitted during the Open-label Period.
  Interventions: Drug: Sebelipase Alfa
- Open-label Placebo/Sebelipase Alfa (Experimental): Participants who were randomized to receive placebo during the Double-blind Period and received sebelipase alfa in the Open-label Period. All participants received sebelipase alfa at a dose of 1 mg/kg qow, irrespective of treatment received in the Double-blind Period. Dose modifications were permitted during the Open-label Period.
  Interventions: Drug: Sebelipase Alfa

INTERVENTIONS:
Drug: Sebelipase Alfa — IV infusions of sebelipase alfa
  Other Names: SBC-102
  Arms: Double-blind Sebelipase Alfa; Open-label Placebo/Sebelipase Alfa; Open-label Sebelipase Alfa/Sebelipase Alfa
Drug: Placebo — IV infusions of matched placebo
  Arms: Double-blind Placebo

SUMMARY:
This Phase 3 study evaluated the efficacy and safety of 1 milligram/kilogram (mg/kg) intravenous (IV) infusions of SBC-102 (sebelipase alfa) administered every other week (qow) in participants with late onset lysosomal acid lipase deficiency (LAL-D) (cholesteryl ester storage disease [CESD]).

Late-onset LAL-D is an underappreciated cause of cirrhosis, liver failure and dyslipidemia. There is currently no standard treatment for LAL-D other than supportive care. Enzyme replacement therapy may be a potential new treatment option for LAL-D participants.

DETAILED DESCRIPTION:
Lysosomal acid lipase deficiency (LAL-D) is a genetic disease characterized by abnormal lipid accumulation in many parts of the body due to a marked decrease in activity of the enzyme lysosomal acid lipase (LAL).

The LAL-D disease spectrum ranges from a presentation in infants that is rapidly progressive to a presentation that occurs in childhood, adolescence, or less frequently, in adulthood in which the rate of disease progression is more variable. Irrespective of where a patient is on the disease spectrum, LAL-D is associated with significant burden of disease and a shortened life expectancy in some patients.

The non-infantile onset form of the disease, also known as CESD, occurs in both children and adults and is an under-appreciated cause of fatty liver with prominent microvesicular steatosis, fibrosis, and cirrhosis. Although the natural history of the disease has not been well studied, serious complications are frequently described, including early death, liver transplantation, or cardiovascular accidents. Other complications include premature atherosclerosis (hardening of arteries) associated with high levels of total cholesterol and low-density lipoprotein (LDL) cholesterol, often called the "bad" cholesterol. The levels of triglycerides can also be high and the levels of high-density lipoprotein (HDL) cholesterol (the "good" cholesterol) are typically low.

In the past, treatments mainly focused on control of the lipid abnormalities through diet and the use of lipid-lowering medications, which only address some aspects of the disease, while progression to fibrosis and cirrhosis may still occur. In preclinical studies and clinical studies in participants with LAL-D, treatment with SBC-102 (sebelipase alfa, Kanuma®) has been shown to produce improvements in markers of liver damage and in the lipid abnormalities. The purpose of this study was to examine the effects of using SBC-102 to treat LAL-D through a placebo-controlled, randomized, double-blinded study in children and adults.

This multicenter, randomized, double-blind, placebo-controlled study involving 66 participants evaluated the safety and efficacy of enzyme-replacement therapy with sebelipase alfa (administered intravenously at a dose of 1 mg/kg of body weight qow). The study included a 20-week placebo-controlled period followed by open-label treatment periods for all participants. The primary end-point was normalization of the alanine aminotransferase level. Secondary end-points included additional disease-related efficacy and safety assessments.

Final study results have not been published in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Participant and/or participant's parent or legal guardian provided informed consent.
* Participant was ≥ 4 years of age on the date of informed consent.
* Deficiency of LAL enzyme activity confirmed by dried blood spot testing at screening.
* Alanine aminotransferase ≥ 1.5x upper limit of normal on 2 consecutive screening measurements obtained at least 1 week apart.
* Female participants of childbearing potential must not have been pregnant or breastfeeding and must have agreed to use a medically acceptable method of preventing contraception from screening until 4 weeks after the last dose of study drug.
* Participant receiving lipid-lowering therapies must have been on a stable dose of the medication for at least 6 weeks prior to randomization and was willing to remain on a stable dose for at least the first 32 weeks of treatment in the study.
* Participant receiving medications for the treatment of nonalcoholic fatty liver disease must have been on a stable dose for at least 16 weeks prior to randomization and was willing to remain on a stable dose for at least the first 32 weeks of treatment in the study.

Exclusion Criteria:

* Severe hepatic dysfunction (Child-Pugh Class C).
* Other medical conditions or comorbidities, which, in the opinion of the Investigator, would have interfered with study compliance or data interpretation.
* Previous hematopoietic or liver transplant procedure.
* Received treatment with high-dose corticosteroids (acute or chronic) within 26 weeks. (Note: Participants receiving maintenance therapy with low-dose oral, intranasal, topical, or inhaled corticosteroids were considered eligible for the study).
* Known hypersensitivity to eggs.
* Participated in a study employing an investigational medicinal product within 4 weeks prior to randomization.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-01-22 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florian Abel, MD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (40):
- United States (11):
  - Tucson, Arizona
  - Palo Alto, California
  - San Francisco, California
  - Wilmington, Delaware
  - Chicago, Illinois
  - Boston, Massachusetts
  - Buffalo, New York
  - Manhasset, New York
  - New York, New York
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
- Córdoba, Argentina
- Australia (4):
  - Brisbane
  - New Lambton
  - Parkville
  - Perth
- Zagreb, Croatia
- Czechia (2):
  - Olomouc
  - Prague
- France (2):
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (3):
  - Freiburg im Breisgau
  - Mainz
  - Munich
- Italy (3):
  - Bergamo
  - Genoa
  - Padua
- Japan (2):
  - Tokyo
  - Tottori
- Mexico City, Mexico
- Warsaw, Poland
- Moscow, Russia
- Spain (3):
  - Elche
  - Madrid
  - Oviedo
- Turkey (Türkiye) (2):
  - Ankara
  - Izmir
- United Kingdom (3):
  - Cambridge
  - London
  - Plymouth

REFERENCES:
- [Background] Wilson DP, Friedman M, Marulkar S, Hamby T, Bruckert E. Sebelipase alfa improves atherogenic biomarkers in adults and children with lysosomal acid lipase deficiency. J Clin Lipidol. 2018 May-Jun;12(3):604-614. doi: 10.1016/j.jacl.2018.02.020. Epub 2018 Mar 9. PMID 29628368
- [Background] Burton BK, Balwani M, Feillet F, Baric I, Burrow TA, Camarena Grande C, Coker M, Consuelo-Sanchez A, Deegan P, Di Rocco M, Enns GM, Erbe R, Ezgu F, Ficicioglu C, Furuya KN, Kane J, Laukaitis C, Mengel E, Neilan EG, Nightingale S, Peters H, Scarpa M, Schwab KO, Smolka V, Valayannopoulos V, Wood M, Goodman Z, Yang Y, Eckert S, Rojas-Caro S, Quinn AG. A Phase 3 Trial of Sebelipase Alfa in Lysosomal Acid Lipase Deficiency. N Engl J Med. 2015 Sep 10;373(11):1010-20. doi: 10.1056/NEJMoa1501365. PMID 26352813
- [Derived] Burton BK, Feillet F, Furuya KN, Marulkar S, Balwani M. Sebelipase alfa in children and adults with lysosomal acid lipase deficiency: Final results of the ARISE study. J Hepatol. 2022 Mar;76(3):577-587. doi: 10.1016/j.jhep.2021.10.026. Epub 2021 Nov 10. PMID 34774639
- [Derived] Valayannopoulos V, Malinova V, Honzik T, Balwani M, Breen C, Deegan PB, Enns GM, Jones SA, Kane JP, Stock EO, Tripuraneni R, Eckert S, Schneider E, Hamilton G, Middleton MS, Sirlin C, Kessler B, Bourdon C, Boyadjiev SA, Sharma R, Twelves C, Whitley CB, Quinn AG. Sebelipase alfa over 52 weeks reduces serum transaminases, liver volume and improves serum lipids in patients with lysosomal acid lipase deficiency. J Hepatol. 2014 Nov;61(5):1135-42. doi: 10.1016/j.jhep.2014.06.022. Epub 2014 Jun 30. PMID 24993530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 study centers located in 17 countries were initiated in this study. Participants were enrolled and treated at 41 centers in 15 countries, including 35 primary centers where participants initiated treatment and 6 qualified local medical centers where participants who were medically stable were transferred for long-term treatment.
Pre-assignment Details: To assess eligibility, participants were screened for a period of up to 6 weeks prior to enrollment in the study. A total of 86 participants were screened. Six of these participants underwent rescreening (of which 2 were eligible for the study). In total, 66 participants were eligible for the study and 20 participants were screen failures.
Groups:
- Double-blind Sebelipase Alfa: Double-blind Period: Intravenous (IV) infusions of sebelipase alfa at a dose of 1 milligram/kilogram (mg/kg) administered every other week (qow).
- Double-blind Placebo: Double-blind Period: IV infusions of placebo administered qow.
- Open-label Sebelipase Alfa/Sebelipase Alfa: Participants who were randomized to receive sebelipase alfa during the Double-blind Period and also received sebelipase alfa in the Open-label Period. All participants received sebelipase alfa at a dose of 1 mg/kg qow, irrespective of treatment received in the Double-blind Period.
- Open-label Placebo/Sebelipase Alfa: Participants who were randomized to receive placebo during the Double-blind Period and received sebelipase alfa in the Open-label Period. All participants received sebelipase alfa at a dose of 1 mg/kg qow, irrespective of treatment received in the Double-blind Period.
Period: Double-blind Period
Arm/Group | Double-blind Sebelipase Alfa | Double-blind Placebo | Open-label Sebelipase Alfa/Sebelipase Alfa | Open-label Placebo/Sebelipase Alfa
Started | 36 | 30 | 0 | 0
Received at Least 1 Dose of Study Drug | 36 | 30 | 0 | 0
Completed | 35 | 30 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Open-label Period
Arm/Group | Double-blind Sebelipase Alfa | Double-blind Placebo | Open-label Sebelipase Alfa/Sebelipase Alfa | Open-label Placebo/Sebelipase Alfa
Started | 0 | 0 | 36 (1 participant who did not complete Double-blind Period due to AE rechallenged for Open-label Period) | 30
Received at Least 1 Dose of Study Drug | 0 | 0 | 36 | 30
Completed | 0 | 0 | 32 | 27
Not Completed | 0 | 0 | 4 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Discontinued by Sponsor | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose (or any portion of a dose) of sebelipase alfa or placebo in the Double-blind Period.
Groups:
- Double-Blind Sebelipase Alfa: Double-blind Period: IV infusions of sebelipase alfa at a dose of 1 mg/kg administered qow.
- Total: Total of all reporting groups
Arm/Group | Double-Blind Sebelipase Alfa | Double-Blind Placebo | Total
Number analyzed (Participants) | 36 | 30 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] — Double-blind Period
  years | 16.9 (11.6) | 15.2 (10.2) | 16.1 (10.9)
Age, Continuous [Mean (Standard Deviation); unit: years] — Open-label Period
  years | 17.39 (11.529) | 15.70 (10.283) | 16.62 (10.930)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 18 | 15 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 30 | 26 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 27 | 28 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants Achieving Alanine Aminotransferase Normalization
Description: Alanine aminotransferase (ALT) normalization was defined as an abnormal baseline value (ALT > the age- and gender-specific upper limit of normal [ULN] provided by the central laboratory performing the assay) that becomes normal (< ULN). Alanine aminotransferase normalization was evaluated at the end of the Double-blind Period (the last double-blind assessment) and at the end of the Open-label Period (last open-label assessment). Baseline for the Open-label Period was defined relative to the first infusion of sebelipase alfa, which occurred at Week 0 for participants in the sebelipase alfa/sebelipase alfa group and Week 22 for participants in the placebo/sebelipase alfa group. The last open-label assessment varied by participant, depending on whether a participant completed treatment through Week 256 or discontinued prior to this timepoint to transition out of clinical study settings.
Time Frame: Double-blind Period: Baseline to the end of the Double-blind Period (Week 20). Open-label Period: Baseline to the last Open-label assessment (up to Week 256)
Population: Double-blind Period: All participants in the Full Analysis Set (defined as participants who received at least 1 dose [or any portion of a dose] of sebelipase alfa or placebo).
  Open-Label Period: All participants in the Extension Set (defined as participants who received at least 1 dose [or any portion of a dose] of sebelipase alfa).
Measure: Number; unit: percentage of participants
Arm/Group | Double-blind Sebelipase Alfa | Double-blind Placebo | Open-label Sebelipase Alfa/Sebelipase Alfa | Open-label Placebo/Sebelipase Alfa
Number analyzed (Participants) | 36 | 30 | 36 | 30
percentage of participants | 31 | 7 | 56 | 37
Statistical Analysis 1: Comparison: Double-blind Sebelipase Alfa vs Double-blind Placebo; A sample size of 50 randomized participants (approximately 25 participants per treatment group) provided 97% power to detect a statistically significant difference between sebelipase alfa and placebo, using Fisher's exact test at α=0.05; Test type: Superiority; p = 0.0271, Fisher Exact; Fisher's exact test at α=0.05

2. Secondary Outcome: Percent Change From Baseline In Low-density Lipoprotein Cholesterol (LDL-C)
Description: Relative reduction (percentage change from baseline) in LDL-C, as assessed by laboratory measurements was evaluated at the end of the Double-blind Period and at the end of the Open-label Period. Baseline for the Open-label Period was defined relative to the first infusion of sebelipase alfa, which occurred at Week 0 for participants in the sebelipase alfa/sebelipase alfa group and Week 22 for participants in the placebo/sebelipase alfa group. The last open-label assessment varied by participant, depending on whether a participant completed treatment through Week 256 or discontinued prior to this timepoint to transition out of clinical study settings.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-blind Sebelipase Alfa | Double-blind Placebo | Open-label Sebelipase Alfa/Sebelipase Alfa | Open-label Placebo/Sebelipase Alfa
Number analyzed (Participants) | 36 | 30 | 36 | 30
percent change | -28.42 (22.304) | -6.25 (13.015) | -19.74 (33.262) | -18.09 (33.685)
Statistical Analysis 1: Comparison: Double-blind Sebelipase Alfa vs Double-blind Placebo; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percent Change From Baseline In Non-high Density Lipoprotein Cholesterol (Non-HDL-C)
Description: Relative reduction (percent change from baseline) in non-HDL-C, as assessed by laboratory measurements, was evaluated at the end of the Double-blind Period and the Open-label Period. Baseline for the Open-label Period was defined relative to the first infusion of sebelipase alfa, which occurred at Week 0 for participants in the sebelipase alfa/sebelipase alfa group and Week 22 for participants in the placebo/sebelipase alfa group. The last open-label assessment varied by participant, depending on whether a participant completed treatment through Week 256 or discontinued prior to this timepoint to transition out of clinical study settings.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind Sebelipase Alfa | Double-Blind Placebo | Open-Label Sebelipase Alfa/Sebelipase Alfa | Open-Label Placebo/Sebelipase Alfa
Number analyzed (Participants) | 36 | 30 | 36 | 30
percent change | -27.97 (18.612) | -6.94 (10.922) | -19.75 (26.875) | -18.34 (29.177)
Statistical Analysis 1: Comparison: Double-Blind Sebelipase Alfa vs Double-Blind Placebo; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percentage Of Participants Achieving Aspartate Aminotransferase Normalization
Description: Aspartate aminotransferase (AST) normalization was defined as an abnormal baseline value (AST > the age- and gender-specific ULN provided by the central laboratory performing the assay) that becomes normal (< ULN). AST normalization was evaluated at the end of the Double-blind Period (the last Double-blind assessment) and at the end of the Open-label Period (last open-label assessment).
  Baseline for the Open-label Period was defined relative to the first infusion of sebelipase alfa, which occurred at Week 0 for participants in the sebelipase alfa/sebelipase alfa group and Week 22 for participants in the placebo/sebelipase alfa group. The last open-label assessment varied by participant, depending on whether a participant completed treatment through Week 256 or discontinued prior to this timepoint to transition out of clinical study settings.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Sebelipase Alfa | Double-Blind Placebo | Open-Label Sebelipase Alfa/Sebelipase Alfa | Open-Label Placebo/Sebelipase Alfa
Number analyzed (Participants) | 36 | 29 | 36 | 29
percentage of participants | 42 | 3 | 69 | 62
Statistical Analysis 1: Comparison: Double-Blind Sebelipase Alfa vs Double-Blind Placebo; Test type: Superiority; p = 0.0003, Fisher Exact

5. Secondary Outcome: Percent Change From Baseline In Triglycerides
Description: Relative reduction (percent change from baseline) in triglycerides, as assessed by laboratory measurements, was evaluated at the end of the Double-blind Period and the Open-label Period. Baseline for the Open-label Period was defined relative to the first infusion of sebelipase alfa, which occurred at Week 0 for participants in the sebelipase alfa/sebelipase alfa group and Week 22 for participants in the placebo/sebelipase alfa group. The last open-label assessment varied by participant, depending on whether a participant completed treatment through Week 256 or discontinued prior to this timepoint to transition out of clinical study settings.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind Sebelipase Alfa | Double-Blind Placebo | Open-Label Sebelipase Alfa/Sebelipase Alfa | Open-Label Placebo/Sebelipase Alfa
Number analyzed (Participants) | 36 | 30 | 36 | 30
percent change | -25.45 (29.411) | -11.14 (28.827) | -11.87 (34.580) | -19.63 (27.066)
Statistical Analysis 1: Comparison: Double-Blind Sebelipase Alfa vs Double-Blind Placebo; Test type: Superiority; p = 0.0375, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percent Change From Baseline In High-density Lipoprotein Cholesterol (HDL-C)
Description: Relative increase (percent change from baseline) in HDL-C, assessed by laboratory measurements, was evaluated at the end of the Double-blind Period and the Open-label Period. Baseline for the Open-label Period was defined relative to the first infusion of sebelipase alfa, which occurred at Week 0 for participants in the sebelipase alfa/sebelipase alfa group and Week 22 for participants in the placebo/sebelipase alfa group. The last open-label assessment varied by participant, depending on whether a participant completed treatment through Week 256 or discontinued prior to this timepoint to transition out of clinical study settings.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind Sebelipase Alfa | Double-Blind Placebo | Open-Label Sebelipase Alfa/Sebelipase Alfa | Open-Label Placebo/Sebelipase Alfa
Number analyzed (Participants) | 36 | 30 | 36 | 30
percent change | 19.57 (16.833) | -0.29 (12.360) | 31.65 (28.971) | 34.78 (29.927)
Statistical Analysis 1: Comparison: Double-Blind Sebelipase Alfa vs Double-Blind Placebo; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percent Change From Baseline In Liver Fat Content
Description: Decrease in liver fat content, as assessed by magnetic resonance imaging (MRI), was evaluated in participants for whom imaging was performed. Baseline for the Open-label Period was defined relative to the first infusion of sebelipase alfa, which occurred at Week 0 for participants in the sebelipase alfa/sebelipase alfa group and Week 22 for participants in the placebo/sebelipase alfa group. The last open-label assessment varied by participant, depending on whether a participant completed treatment through Week 256 or discontinued prior to this timepoint to transition out of clinical study settings.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind Sebelipase Alfa | Double-Blind Placebo | Open-Label Sebelipase Alfa/Sebelipase Alfa | Open-Label Placebo/Sebelipase Alfa
Number analyzed (Participants) | 32 | 25 | 35 | 25
percent change | -31.98 (26.763) | -4.21 (15.559) | -9.89 (32.892) | -0.93 (37.233)
Statistical Analysis 1: Comparison: Double-Blind Sebelipase Alfa vs Double-Blind Placebo; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Participants With Improvement In Liver Histopathology (Decrease Of > 5% In Hepatic Steatosis Score)
Description: The number of participants who had an improvement in hepatic histopathology (defined as a decrease of > 5% in hepatic steatosis score, assessed by morphometry), as determined by blinded central pathologist review, in the participants for whom liver biopsy was performed. Baseline for the Open-label Period was defined relative to the first infusion of sebelipase alfa, which occurred at Week 0 for participants in the sebelipase alfa/sebelipase alfa group and Week 22 for participants in the placebo/sebelipase alfa group.
Time Frame: Double-blind Period: Baseline to the end of the Double-blind Period (Week 20). Open-label Period: Baseline up to Week 52.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Double-Blind Sebelipase Alfa | Double-Blind Placebo | Open-Label Sebelipase Alfa/Sebelipase Alfa | Open-Label Placebo/Sebelipase Alfa
Number analyzed (Participants) | 16 | 10 | 12 | 6
participants | 10 | 4 | 7 | 4
Statistical Analysis 1: Comparison: Double-Blind Sebelipase Alfa vs Double-Blind Placebo; Test type: Superiority; p = 0.4216, Fisher Exact

9. Secondary Outcome: Percent Change From Baseline In Liver Volume
Description: Relative reduction (percent change from baseline) in liver volume, as assessed by MRI, was evaluated in participants for whom imaging was performed. Baseline for the Open-label Period was defined relative to the first infusion of sebelipase alfa, which occurred at Week 0 for participants in the sebelipase alfa/sebelipase alfa group and Week 22 for participants in the placebo/sebelipase alfa group. The last open-label assessment varied by participant, depending on whether a participant completed treatment through Week 256 or discontinued prior to this timepoint to transition out of clinical study settings.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind Sebelipase Alfa | Double-Blind Placebo | Open-Label Sebelipase Alfa/Sebelipase Alfa | Open-Label Placebo/Sebelipase Alfa
Number analyzed (Participants) | 33 | 27 | 36 | 27
percent change | -10.28 (10.510) | -2.66 (10.107) | -24.04 (15.792) | -21.55 (11.727)
Statistical Analysis 1: Comparison: Double-Blind Sebelipase Alfa vs Double-Blind Placebo; Test type: Superiority; p = 0.0068, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: In the Double-blind Period, adverse events were assessed on or after the first infusion of study drug until Week 20. In the Open-label Period, adverse events were assessed after the first infusion of study drug on Week 22 up to Follow-up call (4 weeks [+ 7 days] after the last infusion of sebelipase alfa).
Description: Adverse events were obtained through spontaneous reporting or were elicited by specific questioning of the participant or the participant's parent or legal guardian.
Arm/Group | Double-blind Sebelipase Alfa | Double-blind Placebo | Open-label Sebelipase Alfa/Sebelipase Alfa | Open-label Placebo/Sebelipase Alfa
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/30 | 0/36 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/36 | 1/30 | 6/36 | 5/30
Other Adverse Events (participants affected / at risk) | 31/36 | 28/30 | 35/36 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Sebelipase Alfa (N=36) | Double-blind Placebo (N=30) | Open-label Sebelipase Alfa/Sebelipase Alfa (N=36) | Open-label Placebo/Sebelipase Alfa (N=30)
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1
Infusion-related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — Procedural pain after liver biopsy unrelated to study drug.
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperaemia (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Double-blind Sebelipase Alfa (N=36) | Double-blind Placebo (N=30) | Open-label Sebelipase Alfa/Sebelipase Alfa (N=36) | Open-label Placebo/Sebelipase Alfa (N=30)
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 7 | 11
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 7 | 9
Constipation (Gastrointestinal disorders) | 3 | 1 | 4 | 4
Nausea (Gastrointestinal disorders) | 3 | 2 | 5 | 3
Vomiting (Gastrointestinal disorders) | 3 | 3 | 9 | 7
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 10 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 6 | 10 | 5
Nasopharyngitis (Infections and infestations) | 4 | 3 | 17 | 14
Rhinitis (Infections and infestations) | 2 | 3 | 4 | 9
Sinusitis (Infections and infestations) | 2 | 0 | 4 | 0
Tonsillitis (Infections and infestations) | 2 | 4 | 4 | 3
Pharyngitis (Infections and infestations) | 0 | 5 | 6 | 5
Respiratory tract infection viral (Infections and infestations) | 0 | 2 | 0 | 4
Varicella (Infections and infestations) | 0 | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 5 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 12 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 8 | 5
Pyrexia (General disorders) | 7 | 6 | 15 | 9
Asthenia (General disorders) | 3 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 3 | 3
Vaccination site pain (General disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 10 | 6 | 19 | 12
Syncope (Nervous system disorders) | 2 | 0 | 1 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 1 — Procedural pain after liver biopsy deemed by the Investigator to be unrelated to study drug.
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 4
Body temperature increased (Investigations) | 2 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 4
Anxiety (Psychiatric disorders) | 2 | 0 | 2 | 1
Arrhythmia (Cardiac disorders) | 0 | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 5
Gastroenteritis (Infections and infestations) | 1 | 0 | 5 | 7
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 3
Influenza (Infections and infestations) | 0 | 1 | 3 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 3
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 3
Vulvovaginitis (Infections and infestations) | 0/18 | 0/15 | 1/18 | 2/15 — Adverse event occurring in female participants only.
Otitis media (Infections and infestations) | 0 | 0 | 3 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 2
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 2
Ear infection (Infections and infestations) | 0 | 0 | 2 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 6 | 3
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 4
Malaise (General disorders) | 0 | 1 | 2 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 4 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0/18 | 1/15 | 3/18 | 4/15 — Adverse event occurring in female participants only.
Blood cholesterol increased (Investigations) | 0 | 0 | 2 | 0
Blood pressure increased (Investigations) | 0 | 0 | 2 | 0
Cardiac murmur (Investigations) | 0 | 0 | 2 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 8 | 4
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 4 | 2
Autism spectrum disorder (Psychiatric disorders) | 0 | 0 | 2 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 1 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator may publish or make an individual oral or written presentation of publication of study results either 1) after Alexion publishes the study data or 2) 18 months after the completion of the study, whichever comes first.

Alexion reserves the right to review and comment on a communication at least 30 days prior to submission with a provision to extend the review for an additional 60 days where information is relevant to a patent application.